CLINICAL TRIAL: NCT00010218
Title: Phase II Trial Of Karenitecin (IND 57250) In Patients With Relapsed or Refractory Non-small Cell Lung Cancer
Brief Title: Karenitecin in Treating Patients With Relapsed or Refractory Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30004; U10CA031946 (NIH); CLB-30004; CDR0000068456 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — cositecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- karenitecin (Experimental): Patients receive karenitecin IV over 60 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease after 6 courses may receive 2 additional courses beyond best response.
  Patients are followed every 3 months for 1 year and then every 6 months thereafter.
  Interventions: Drug: karenitecin

INTERVENTIONS:
Drug: karenitecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of karenitecin in treating patients who have relapsed or refractory non-small cell lung cancer

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response in patients with relapsed or refractory non-small cell lung cancer treated with karenitecin as salvage chemotherapy.
* Determine the effect of prior response to chemotherapy on response to this drug in these patients.
* Determine survival and failure-free survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: Patients are stratified according to response to prior chemotherapy (relapsed vs refractory).

Patients receive karenitecin IV over 60 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease after 6 courses may receive 2 additional courses beyond best response.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

PROJECTED ACCRUAL: A minimum of 45 patients (25 for stratum I and 20 for stratum II) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed relapsed or refractory non-small cell lung carcinoma (NSCLC)

  * Squamous cell carcinoma
  * Basaloid carcinoma
  * Adenocarcinoma
  * Bronchoalveolar carcinoma
  * Adenosquamous cell carcinoma
  * Large cell carcinoma
  * Large cell neuroendocrine carcinoma
  * Giant cell carcinoma
  * Sarcomatoid carcinoma
  * Non-small cell carcinoma not otherwise specified
* Histologic or cytologic documentation of recurrence required if disease previously completely resected
* Must have had only 1 prior chemotherapy regimen, including adjuvant or neoadjuvant therapy for NSCLC
* At least 1 unidimensionally measurable lesion

  * At least 20 mm with conventional techniques OR
  * At least 10 mm with spiral CT scan
  * Lesions that are not considered measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions in a previously irradiated area
* Controlled CNS metastases allowed if patient is neurologically stable and off steroids

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than upper limit of normal

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin)
* No prior irinotecan or other camptothecin drug
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* No concurrent hormonal therapy except for non-cancer-related conditions (e.g., insulin for diabetes)
* No concurrent steroids except for adrenal failure

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy for symptomatic lesions or those that might produce disability (e.g., painful bone metastases) allowed if other measurable disease present
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2001-04; Primary Completion 2003-04 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (44):
- United States (44):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Miller AA, Herndon JE 2nd, Gu L, Green MR; Cancer and Leukemia Group B. Phase II trial of karenitecin in patients with relapsed or refractory non-small cell lung cancer (CALGB 30004). Lung Cancer. 2005 Jun;48(3):399-407. doi: 10.1016/j.lungcan.2004.11.019. Epub 2005 Jan 23. PMID 15893009
- [Result] Herndon JE, Miller AA, Zhang C, et al.: Phase II trial of karenitecin in patients with refractory non-small cell lung cancer (NSCLC): CALGB 30004 . [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2706, 673, 2003.